CLINICAL TRIAL: NCT00761514
Title: Evaluation of Quality of Life Changes in Puerto Rican Subjects With Active Rheumatoid Arthritis Treated With Humira as Their First Anti-TNF Monoclonal Antibody (VIVIR)
Brief Title: Evaluation of Quality of Life Changes in Puerto Rican Subjects With Active Rheumatoid Arthritis Treated With Humira
Acronym: VIVIR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated due to low enrollment.
Sponsor: Abbott (Industry)
Responsible Party: Carlos R. Rivera-Vázquez, MD/Medical Director, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W06-407
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Results first posted 2009-11-19 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): All subjects will receive Adalimumab
  Interventions: Drug: Humira (adalimumab)

INTERVENTIONS:
Drug: Humira (adalimumab) — 40 mg eow
  Other Names: ABT-D2E7; adalimumab; Humira

SUMMARY:
The primary objective of this study is to evaluate quality of life changes in Puerto Rican subjects with Rheumatoid Arthritis treated with Humira (adalimumab) as their first Anti-TNF Monoclonal Antibody.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to any study-specific procedures.
* Subject is 18 years of age or older.
* If female, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing one of the following methods of birth control:

  * condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD).
  * contraceptives (oral or parenteral) for three months prior to study drug administration).
  * a vasectomized partner.
  * total abstinence from sexual intercourse.
* If female, the results of a serum pregnancy test performed at Screening, prior to the first dose of Humira (adalimumab) must be negative.
* Subject has confirmed diagnosis of active rheumatoid arthritis as defined by >= 6 swollen joints and >= 9 tender joints.
* Subject has an Erythrocyte Sedimentation Rate (ESR) of > 20 mm/hr. ESR will be measured using the Westergren method.
* Subject meets the American College of Rheumatology (ACR) criteria for diagnosis of rheumatoid arthritis (RA) for at least 3 months prior to enrollment and requires to be started in a biologic containing treatment for the first time, and the investigator chooses Humira (adalimumab).
* Subject has had unsatisfactory response or intolerance to one or more prior disease-modifying antirheumatic drugs (DMARDS) (e.g., hydroxychloroquine, leflunomide, methotrexate, parenteral gold, sulfasalazine, azathioprine or any combination of those).
* Subject will have an evaluation for latent tuberculosis with a tuberculosis (TB) skin test done in the screening visit. Subjects who have evidence of prior TB infection should be given prophylaxis in accordance with Centers for Disease Control and Prevention (CDC) guidelines.

Exclusion Criteria:

* Subjects who have had prior treatment with cyclophosphamide, chlorambucil or any other Tumor Necrosis Factor (TNF) biologic as etanercept, infliximab, anakinra, abatacept and adalimumab.
* Subjects who have been previously treated with total lymphoid irradiation or anti-CD4 or CAMPATH 1H monoclonal antibodies resulting in persistent CD4 lymphopenia (CD4 lymphocytes <= 500/mm3).
* Subject has had prior treatment with intravenous (IV) immunoglobulin or any investigational agent within 30 days of screening visit.
* Subject has a history of cancer within the past 10 years other than resected basal cell or squamous cell carcinomas of the skin.
* Subject has a history of malignant lymphoma or leukemia regardless of time since diagnosis.
* Subject has a history of or current acute inflammatory joint disease of origin other than RA, e.g., Mixed Connective Tissue Disease (MCTD), Systematic Lupus Erythematosus (SLE), etc.
* Subject has a history of uncontrolled diabetes mellitis, unstable ischemic heart disease, active inflammatory bowel disease, active peptic ulcer disease, recent cerebrovascular accident (CVA) (within 3 months) which, in the opinion of the investigator, would put the subject at risk by participation in the protocol.
* Subject has a history of active tuberculosis or listeriosis, or other active infections suggestive of significant or profound immunosuppression, such as Pneumocystis carinii, aspergillosis or other systemic protozoan or fungal infections.
* Subject has a positive serology for Hepatitis B or Hepatitis C indicating active infection.
* Subject has a history of positive HIV status defined by an enzyme-linked immunosorbent assay (ELISA) positive test confirmed by a Western blot test and/or polymerase chain reaction (PCR).
* Subject has had a persistent or severe infection(s) requiring hospitalization or treatment with intravenous (IV) antibiotics within 30 days, or oral antibiotics within 14 days, prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos R. Rivera-Vàzquez, MD, Study Director — Abbott
Locations (9):
- Puerto Rico (9):
  - Aguada
  - Bayamón
  - AJP Med, Inc. PSA, Caguas
  - Caguas
  - Humacao
  - Manatí
  - Rio Piedras
  - San Juan Arthritis & Research Center, San Juan
  - San Juan

REFERENCES:
- See also: Link to product information — http://www.humira.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 10 study sites in Puerto Rico beginning in November 2006.
Pre-assignment Details: Not applicable. This was an open-label study. All enrolled subjects received treatment.
Groups:
- Open-label Treatment With 40 mg Adalimumab Every Other Week: All subjects received 40 mg Adalimumab by subcutaneous injection every other week for up to 24 weeks.
Period: Overall Study
Arm/Group | Open-label Treatment With 40 mg Adalimumab Every Other Week
Started | 14
Completed | 7
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Health insurance didn't cover study drug | 1
Not completed — Problem complying with study visit | 1
Not completed — Unable to pay for medications | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Treatment With 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 61.29 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 14

OUTCOME MEASURES:

1. Secondary Outcome: Percent Change From Baseline to Week 24 in Average Score on the Short Disease Activity Score
Description: On visual analog scale (VAS), patient marks activity of rheumatoid arthritis in previous 24 hours (0 mm=no symptoms; 100 mm=very active). On another VAS, patient marks how much pain (0 mm=no pain; 100 mm=severe pain) he/she had because of the illness in previous week. Patient also marks tender joints and swollen joints on body diagrams. Number of swollen and painful joints and values on VAS are used with erythrocyte sedimentation rate to calculate the patient's global assessment of disease activity. High score indicates high activity.
Time Frame: Week 24 of treatment
Population: Available subject data were used in calculations. Missing data were not imputed.
Measure: Number; unit: Percent change in average score
Groups:
- Open-label Treatment With Adalimumab 40 mg Every Other Week: All subjects received 40 mg adalimumab by subcutaneous injection every other week for up to 24 weeks.
Arm/Group | Open-label Treatment With Adalimumab 40 mg Every Other Week
Number analyzed (Participants) | 14
Percent change in average score | 31

2. Primary Outcome: Percent Change From Baseline to Week 24 in Average Score on Section 1 of the Modified Multi-Dimensional Health Assessment Questionnaire (mHAQ) That Includes Ratings of Sleep, Anxiety, Depression or Feeling Blue, and Ability to do Daily Activities.
Description: Section 1 of the mHAQ includes subject ratings of difficulty in: dressing; getting out of bed; lifting a full glass to the mouth; walking outdoors on flat ground; bathing; bending to pick up clothes from floor; getting in/out of car, bus, train, plane; walking 2 miles; participating in sports and games; getting a good night's sleep; dealing with feelings of anxiety, being nervous; dealing with feelings of depression, feeling blue. Without any difficulty=0, With some difficulty=1, With much difficulty=2, Unable to do=3. Ratings are summed. The maximum total score is 39. Low total score is good.
Time Frame: Week 24 of treatment
Population: Available subject data were used in calculations; 14 at Baseline and 7 at Week 24. Missing data were not imputed.
Measure: Number; unit: Percent change in average total score
Arm/Group | Open-label Treatment With Adalimumab 40 mg Every Other Week
Number analyzed (Participants) | 14
Percent change in average total score | 59

ADVERSE EVENTS:
Arm/Group | Open-label Treatment With 40 mg Adalimumab Every Other Week
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Treatment With 40 mg Adalimumab Every Other Week (N=14)
Oropharyngeal herpes simplex pharyngitis (Infections and infestations) | 1
Hospitalization due to fall (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Treatment With 40 mg Adalimumab Every Other Week (N=14)
Erythema surrounding area of Humira injection (Skin and subcutaneous tissue disorders) | 1
Erythema versicular rash (Skin and subcutaneous tissue disorders) | 1
Erythema rash (Skin and subcutaneous tissue disorders) | 1
Fever (Infections and infestations) | 1
Cellulitis right thigh (Skin and subcutaneous tissue disorders) | 1
Sore throat (Infections and infestations) | 1
Epigastric pain (Gastrointestinal disorders) | 1
Non-pruritic areas of erythema on arms (Skin and subcutaneous tissue disorders) | 1
Nasal congestion (General disorders) | 1
Dry mouth (General disorders) | 1
Hair loss (General disorders) | 1
Dry eyes (Eye disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Non-painful purplish spots on arms (Skin and subcutaneous tissue disorders) | 1
High blood pressure (Cardiac disorders) | 1
Lumbar pain (General disorders) | 1
Elevated blood pressure (Cardiac disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Rash on arms and whole body (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
This study was terminated early due to lack of enrollment. Only 7 subjects completed 24 weeks of treatment. That number is too small to provide reliable data on the effectiveness of the treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall provide Abbott at least sixty (60) days prior to publication or presentation, with a draft of the same for Abbott's review and comment, to ascertain whether any patentable subject matter or Abbott confidential infromariont are disclosed therin. Abbott shall return comment within sixty (60) days after receipt of the draft.